CLINICAL TRIAL: NCT07400666
Title: Intra-gastrointestinal Monitoring Device (PressureDOT®) and Centurion Intra-abdominal Pressure Monitoring Device Comparison Study: Pivotal Study of Safety and Performance.
Brief Title: Intra-gastrointestinal Monitoring Device (PressureDOT®) and Centurion IAP Monitoring Device Comparison Study: Pivotal Study of Safety and Performance.
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Dotspace Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: PDT-02-012 V.2025-A.05
Record Dates: First submitted 2026-02-03; First posted 2026-02-10 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Intra Abdominal Pressure; Intra-Abdominal Hypertension
Keywords: comparison study; Digital capsule
MeSH Terms: conditions — Intra-Abdominal Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- ICU patients who require IAP monitoring (Experimental): The subject will have PressureDOT and Centurion IAP monitoring device to collect the IAP data at the same time in the study until the excretion of digital capsule.
  Interventions: Device: digital capsule

INTERVENTIONS:
Device: digital capsule — A digital capsule to monitor intra-gastrointestinal pressure and wirelessly transmit the data to bedside reader for healthcare providers.

SUMMARY:
The proposed clinical study protocol is intended to establish the safety, utility, and reliability of using a pressure-sensing capsule present in a patient's gastrointestinal tract for monitoring intraabdominal pressure (IAP). Monitoring IAP in critically ill patients is common in patients admitted to the ICU following a wide variety of surgical interventions. It has been reported that approximately 50% of critically ill patients will develop intraabdominal hypertension (IAH; defined as an IAP >12 mmHg) while in the ICU, which can be life-threatening due to complications resulting from organ dysfunction, organ failure, impaired ventilation and hemodynamic instability. When IAH is persistent and elevated above 20 mmHg the condition is identified as "Abdominal Compartment Syndrome (ACS)", which necessitates close monitoring of patients with IAH in order to reduce the development of ACS. IAP measurements based on technologies employing the bladder, gastric, inferior vena cava, rectal, vaginal and direct intraperitoneal placements have been reported for assessing IAP. However, the gold standard method for monitoring IAP is the use of an intravesical (bladder) Foley catheter manometric technique. PressureDOT® (Dotspace Inc.) is the investigational pressure-sensing capsule that will be assessed in a parallel device clinical study protocol performed in the same patient.

ELIGIBILITY:
Inclusion Criteria:

1. Patients admitted to the ICU who require IAP monitoring.
2. Are at least 22 years old.
3. Have a BMI greater than 18.5 kg/m², but less than 35 kg/m².
4. Expected survival of at least 5 days.
5. Blood sodium > 130 and < 150 mmol/L.
6. Are able to speak and read English.
7. Have signed an Informed Consent or their legal representative/surrogate has signed an Informed Consent.

Exclusion Criteria:

1. The patient is anticipated to undergo an MRI examination within seven days after ingestion of the capsule.
2. The patient is anticipated to undergo radiotherapy within seven days after ingestion of the capsule.
3. Patients who are on ECMO treatment.
4. Conscious patients with a history of difficulty with swallowing due to functional or anatomic disorder.
5. Patients with a history of bowel stenosis.
6. Patients with a history of bowel mechanical obstruction.
7. Patients with a past history of intestinal diverticula, intestinal obstruction/stenosis, intestinal reconstructed operation or any past history indicating a high risk for capsule retention based on the PI's evaluation and judgement.
8. Patients with obvious clinical evidence of gastrointestinal tract obstruction or severe paralytic ileus that need immediate surgical intervention.
9. Female subjects who are pregnant, planning on becoming pregnant or nursing. To exclude the possibility of pregnancy risk in the enrollment stage, a pregnancy test will be prescribed to the female subjects who fits the fertility status.
10. The presence of any other active implanted device, such as a cardiac pacemaker or other implanted electromedical devices.
11. The presence of any other wireless sensor or transmitter located in the abdomen (excluding compatible devices also in use for pressure sensing within the body).
12. Patients with Crohn's disease or diverticulitis.
13. Patients diagnosed with radiation enteritis.
14. Patients with severe systemic diseases and not allowed to join this study by the principal investor's judgement, such as severe congestive heart failure, renal failure or liver diseases.
15. Congenital anomalies of gastrointestinal tract or any other anatomical abnormality of the head, neck, chest, or abdomen that would be a contraindication to placement of the PressureDOT® device and usage of the external device.
16. Has a BMI > 35 kg/m² or <18.5 kg/m²
17. Subjects with any contraindication to urinary bladder catheterization or intravesical intra-abdominal pressure measurement, including but not limit:

    1. Known or suspected urethral injury, severe urethral stricture or recent pelvic or lower urinary tract trauma.
    2. Recent urological surgery involving the bladder, prostate, or urethra that precludes safe Foley catheter placement.
    3. Clinically diagnosed urosepsis or active, symptomatic urinary tract infection.
    4. Neurogenic bladder with documented poor bladder compliance, in the judgment of the Principal Investigator.
    5. Confirmed anuria or urinary obstruction that may compromise the accuracy or safety of intravesical pressure measurement.
    6. Gross hematuria or bladder outlet obstruction that contraindicates Foley catheterization.
18. A patient who, in the judgment of the Principal Investigator, is not appropriate for enrollment.
19. A patient or his/her legal representative/surrogate who isn't fluent in English.
20. A patient or his/her legal representative/surrogate who doesn't sign the Informed Consent.

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Estimated)
Dates: Start 2026-07-01 (Estimated); Primary Completion 2026-10-30 (Estimated); Study Completion 2026-11-30 (Estimated)

PRIMARY OUTCOMES:
Number of participants with treatment-related adverse events as assessed by Clavien-Dindo grade. | From deployment of the PressureDOT digital capsule to the 7 days after the digital capsule excretion.
The agreements of two IAP measurement devices. | From the deployment of the PressureDOT digital capsule to 7 days after the digital capsule excretion.
The average time to excrete the PressureDOT digital capsule in the enrolled study participants. | From the deployment of the PressureDOT digital capsule to 7 days after the digital capsule excretion.

IPD SHARING:
Plan to Share IPD: Undecided
We will discuss with the clinical sites and PIs for the next steps.